CLINICAL TRIAL: NCT05646602
Title: Impact of Focused Low-intensity Shockwave Therapy (LiSWT) in Penile Disorders (Peyronie's Disease, Erectile Dysfunction, or Both), With or Without Intralesional Clostridial Collagenase (Xiaflex) Injection, Compared With Radial Shock Wave Therapy or Xiaflex Therapy
Brief Title: Focused Shock Wave Therapy Outcomes in Peyronie's Disease and Erectile Dysfunction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Tobias S. Kohler, MD, MPH, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-001663
Record Dates: First submitted 2022-12-02; First posted 2022-12-12 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Peyronie Disease; Penile Curvature; Erectile Dysfunction
MeSH Terms: conditions — Penile Induration; Erectile Dysfunction | interventions — Microbial Collagenase

STUDY DESIGN:
Intervention Model Description: Following enrollment men will be randomized based on the severity of their penile curvature. Separate randomization tables will be established for men with penile curvature (i) 30 to < 60 degrees and (ii) 60-90 degrees. Patients will be randomized in a 1:1 ratio to CCH + LiSWT versus CCH alone within each severity cohort, with the intention to enroll a similar number of patients within each severity group
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Collagenase Clostridium Histolyticum with LiSWT for PD Group (Experimental): Subjects being treated for Peyronie's disease (PD) will have Collagenase Clostridium Histolyticum (CCH) intralesional injection with focused low-intensity shockwave therapy (LiSWT).
  Interventions: Drug: Collagenase Clostridium Histolyticum; Device: Duolith SD1 T-TOP
- Collagenase Clostridium Histolyticum for PD Group (Active Comparator): Subjects being treated for Peyronie's disease (PD) will have Collagenase Clostridium Histolyticum (CCH) intralesional injection
  Interventions: Drug: Collagenase Clostridium Histolyticum
- Radial Shockwave Therapy for ED Group (Active Comparator): Subjects being treated for erectile dysfunction (ED) will have radial shockwave therapy.
  Interventions: Device: Duolith SD1 T-TOP
- Linear Shockwave Therapy for ED Group (Experimental): Subjects being treated for erectile dysfunction (ED) will have linear shockwave therapy
  Interventions: Device: Duolith SD1 T-TOP

INTERVENTIONS:
Drug: Collagenase Clostridium Histolyticum — Intralesional injection
  Other Names: Xiaflex
  Arms: Collagenase Clostridium Histolyticum for PD Group; Collagenase Clostridium Histolyticum with LiSWT for PD Group
Device: Duolith SD1 T-TOP — Delivers low-intensity shockwave therapy, six sessions (once/week) of 2000 shockwaves per session with a constant energy flux density of 0.29 mJ/mm2 and frequency of 3 Hz
  Arms: Collagenase Clostridium Histolyticum with LiSWT for PD Group; Linear Shockwave Therapy for ED Group; Radial Shockwave Therapy for ED Group

SUMMARY:
The purpose of this research is to determine the pure or additional effects of penile shockwave therapy with low intensity linear shock wave machine for penile curvature (and/or erectile dysfunction) vs patients' undergoing other treatments (including Xiaflex therapy, patients that have undergone older generations of SWT, or medical treatment).

ELIGIBILITY:
Inclusion Criteria:

* Peyronie's Disease (PD) at any stage
* The presence of penile plaque or pain at erection or curvature
* PD therapy with or without simultaneous intralesional Xiaflex injection.

Exclusion Criteria:

* Prior penile surgery or LiSWT.
* Erective Dysfunction (ED) not responding to phosphodiesterase-type five inhibitors or intracavernosal injections.
* Unwillingness or inability to provide informed consent.
* Having active or life-threatening coagulopathies ore using anti-coagulation /anti-platelet medications

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in penile curvature | Baseline, 10 weeks
  Measured with a goniometer after artificial erection reported in degree unit of measurements

SECONDARY OUTCOMES:
Change in Sexual function | Baseline, 10 weeks
  Measured using the Sexual Encounter Profile (SEP) questions 2 and 3 to assess functional outcomes on a scale of 0=no sexual activity/did not attempt intercourse; 1=almost never/never; 2=A few times (much less than half the time); 3=Sometimes (about half the time); 4=Most times (much more than half the time); 5=Almost always/always
Change in penile length | Baseline, 10 weeks
Li-SWL related pain at therapy sessions | 6 weeks
  Measured using a visual analog scale (VAS) ranging from 0 (no pain) to 10 (intolerable pain)

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Kohler, MD, MPH, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials